CLINICAL TRIAL: NCT00612911
Title: Cell Therapy in Dilated Cardiomyopathy: A Safety and Feasibility Study Using Autologous Bone Marrow Mononuclear Cells
Brief Title: Cell Therapy in Dilated Cardiomyopathy: Observational Study
Status: Terminated | Type: Observational
Why Stopped: finish study as protocol
Sponsor: Ministry of Health, Brazil (Other Government)
Responsible Party: Helena Martino, Brazil: National Institute of Cardioloy
Other Study IDs: CTDil-1
Record Dates: First submitted 2008-01-23; First posted 2008-02-12 (Estimated); Last update posted 2008-02-12 (Estimated); Status verified 2008-01

CONDITIONS: Cardiomyopathy, Dilated
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Major group: Patients with Idiopathic dilated cardiomyopathy
  Interventions: Other: Cell therapy

INTERVENTIONS:
Other: Cell therapy — bone marrow mononuclear cell

SUMMARY:
Using bone marrow mononuclear cell in 24 patients with Idiopathic dilated cardiomyopathy

DETAILED DESCRIPTION:
Patients with Idiopathic dilated cardiomyopathy class II to IV NYHA with ejection fraction <35% were selected for phase I clinical trial of bone marrow mononuclear cell delivery in the coronary arteries and followed for 6 months

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic dilated cardiomyopathy
* Optimized therapy and for idiopathic dilated cardiomyopathy
* Left ventricular ejection fraction (Simpson) < 35%
* Peak oxygen consumption (VO2 peak) < 16 mL.kg-1min-1
* Functional classes II-IV of the NYHA

Exclusion Criteria:

* dilated cardiopathies of ischemic or chagasic origin
* primary valve disease
* excessive use of alcohol or illicit drugs
* pregnancy
* ventricular arrhythmias
* any co-morbidity with impact on survival

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with idiopathic dilated cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2005-02; Primary Completion 2006-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
echocardiography | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Helena F Martino, Principal Investigator — Brazil: National Insittute of Cardiology
Locations (1):
- INCL - National Institute of Cardiology Laranjeiras, Rio de Janeiro, Rio de Janeiro, Brazil